CLINICAL TRIAL: NCT03150589
Title: A Phase III Randomised, Double-masked, Parallel Group, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics and Immunogenicity Between SB11 and Lucentis® in Subjects With Neovascular Age-related Macular Degeneration
Brief Title: A Study to Compare SB11 (Proposed Ranibizumab Biosimilar) to Lucentis in Subjects With Neovascular Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB11-G31-AMD
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-04

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SB11 (Proposed ranibizumab biosimilar) (Experimental)
  Interventions: Drug: SB11 (Proposed ranibizumab biosimilar)
- Lucentis (ranibizumab) (Active Comparator)
  Interventions: Drug: Lucentis (ranibizumab)

INTERVENTIONS:
Drug: SB11 (Proposed ranibizumab biosimilar) — SB11 (proposed ranibizumab biosimilar) 0.5mg via intravitreal injection every 4 weeks
  Arms: SB11 (Proposed ranibizumab biosimilar)
Drug: Lucentis (ranibizumab) — Lucentis (ranibizumab) 0.5mg via intravitreal injection every 4 weeks
  Arms: Lucentis (ranibizumab)

SUMMARY:
This is a randomised, double-masked, parallel group, multicentre study to evaluate the efficacy, safety, pharmacokinetics and immunogenicity of SB11 compared to Lucentis® in subjects with neovascular AMD.

DETAILED DESCRIPTION:
Subjects will be randomised in a 1:1 ratio to receive either SB11 or Lucentis® (administered via intravitreal (ITV) 0.5 mg every 4 weeks). Investigational Products (IP) (SB11 or Lucentis®) will be administered up to Week 48, and the last assessment will be done at Week 52.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years
2. Newly diagnosed, active subfoveal choroid neovascularisation (CNV) lesion secondary to AMD in the study eye
3. BCVA of 20/40 to 20/200 in the study eye
4. Written informed consent form

Exclusion Criteria:

1. Any previous ITV anti-vascular endothelial growth factor (anti-VEGF) treatment to treat neovascular AMD in either eye
2. Presence of CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, multifocal choroiditis, angioid streaks, history of choroidal rupture or pathologic myopia
3. Any concurrent macular abnormality other than AMD in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Se Joon Woo, Principal Investigator — Seoul National University Bundang Hospital, South Korea
Locations (75):
- United States (19):
  - Retina consultants San Diego, Poway, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Retina Consultants, Fort Myers, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Raj K. Maturi, MD, PC, Indianapolis, Indiana
  - Retina Center of New Jersey, LLC, Bloomfield, New Jersey
  - NJ Retina, Toms River, New Jersey
  - LIVR, Great Neck, New York
  - Long Island Vitreoretinal Consultants, Hauppauge, New York
  - Retina Associates of Western NY, Rochester, New York
  - Retina Vitreous Surgeons fo Central NY, PC, Syracuse, New York
  - Retina Associates of Cleveland, Middleburg Heights, Ohio
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Restina Associates, Austin, Texas
  - Retina consultants of Houston, Conroe, Texas
  - Retina Consultants of Houston, Houston, Texas
- Czechia (6):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hopsital Ostrava, Ostrava
  - Axon Clinical s.r.o., Prague
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- Germany (10):
  - Augenärzte am St. Franziskus-Hospital Münster, Münster, Munster
  - Charite, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Uni Düsseldorf, Düsseldorf
  - University Medical Center, Freiburg, Freiburg im Breisgau
  - Uni Göttingen, Goettigen
  - TU Munich, München
  - MVZ ADTC Siegburg GmbH, Siegburg
  - University of Tuebingen STZ eyetrial at the Department of Ophthalmology, Tübingen
- Hungary (10):
  - Ganglion Orvosi Kozpont, Pécs, Pecs
  - Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Budapest Retina Associates Ltd., Budapest
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Peterfy Sandor utcai Korhaz-Rendelointezet es Baleseti Kozpont, Budapest
  - Semmelweis Egyetem Szemeszeti Klinika, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Szemklinika, Debrecen
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- India (6):
  - Medilink Hospital, Ahmedabad
  - PGIMER, Chandigarh
  - Shankara Netralaya, Chennai
  - Aravind Eye Hospital, Coimbatore
  - Shroff eye Hospital, Mumbai
  - Regional Institute of Opthalmology, Trivandrum
- Poland (7):
  - Centrum Medyczne UNO-MED., Tarnów, Tarnow
  - Szpital Specjalistyczny im Sokołowskiego Oddzial Okulistyczny, Wałbrzych, Walbrzych
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego, Klinika Okulistyki, Wroclaw, Wroclaw
  - Oftalmika ul. Modrzewiowa 15 85-631 Bydgoszcz, Bydgoszcz
  - Specjalistyczna Praktyka Lekarska Prof. E. Wylęgała, Katowice
  - Centrum Medyczne UNO-MED., Krakow
  - Centrum Diagnostyki i Mikrochirurgii Oka LENS, Olsztyn
- Russia (6):
  - "State Autonomous Iinstitution of Healthcare "Republican clinical ophthalmological hospital of MoH of Republic of Tatarstan", Kazan'
  - Deputy Director of The S.N.Fyodorov Eye Microsurgery State Institution Complex, Moscow
  - Federal State Budget Scientific Institution "Scientific Research Institute of Eye Diseases", Moscow
  - Federal State Autonomous Institution "Intersectoral research and technical complex "Eye Microsurgery" named after acad. S.N. Fyodorov" of Ministry of Health of Russian Federation, Novosibirsk
  - Federal State Educational Institution of High Professional Education "1st Saint-Petersburg State Medical University n.a. academic I.P. Pavlov" of Ministry of Healthcare of Russian Federation, Saint Petersburg
  - SBEI HPE "Samara State Medical University" of the MoH of the RF, Samara
- South Korea (7):
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- United Kingdom (4):
  - Queens University Belfast, Belfast
  - Bristol Eye Hospital, Bristol
  - Frimley Park Hospital, Frimley
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bressler NM, Kim T, Oh I, Russo P, Kim MY, Woo SJ. Immunogenicity With Ranibizumab Biosimilar SB11 (Byooviz) and Reference Product Lucentis and Association With Efficacy, Safety, and Pharmacokinetics: A Post Hoc Analysis of a Phase 3 Randomized Clinical Trial. JAMA Ophthalmol. 2023 Feb 1;141(2):117-127. doi: 10.1001/jamaophthalmol.2022.5403. PMID 36520462
- [Derived] Woo SJ, Veith M, Hamouz J, Ernest J, Zalewski D, Studnicka J, Vajas A, Papp A, Gabor V, Luu J, Matuskova V, Yoon YH, Pregun T, Kim T, Shin D, Bressler NM. Efficacy and Safety of a Proposed Ranibizumab Biosimilar Product vs a Reference Ranibizumab Product for Patients With Neovascular Age-Related Macular Degeneration: A Randomized Clinical Trial. JAMA Ophthalmol. 2021 Jan 1;139(1):68-76. doi: 10.1001/jamaophthalmol.2020.5053. PMID 33211076

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SB11 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Started | 351 | 354
Completed | 307 | 327
Not Completed | 44 | 27
Not completed — Withdrawal by Subject | 16 | 9
Not completed — Adverse Event | 7 | 6
Not completed — Protocol Violation | 4 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Death | 2 | 3
Not completed — IP non-compliance and other reasons | 12 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB11 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab) | Total
Number analyzed (Participants) | 351 | 354 | 705
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (8.00) | 73.8 (8.92) | 74.1 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 201 | 403
  Male | 149 | 153 | 302
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 51 | 52 | 103
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 297 | 300 | 597
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA)
Description: The VA was assessed using original series ETDRS charts or 2702 series number charts.
Time Frame: Baseline and Week 8
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | SB11 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 346 | 348
letters | 6.26 (0.51) | 7.08 (0.51)

2. Primary Outcome: Change From Baseline in Central Subfield Thickness (CST)
Description: The average retinal thickness in the central 1-mm area in the ETDRS grid (CST) was evaluated using (Optical Coherence Tomography) OCT
Time Frame: Baseline and Week 4
Population: Per-Protocol Set for CST
Measure: Least Squares Mean (Standard Error); unit: μm
Arm/Group | SB11 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
Number analyzed (Participants) | 342 | 338
μm | -108.40 (4.65) | -100.05 (4.64)

ADVERSE EVENTS:
Time Frame: From the time the subject signed the written informed consent until Week 52 (EOS Visit) or ET Visit
Description: All AEs (ocular or non-ocular) were recorded.
Arm/Group | SB11 (Proposed Ranibizumab Biosimilar) | Lucentis (Ranibizumab)
All-Cause Mortality (participants affected / at risk) | 0/350 | 0/354
Serious Adverse Events (participants affected / at risk) | 52/350 | 52/354
Other Adverse Events (participants affected / at risk) | 111/350 | 126/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB11 (Proposed Ranibizumab Biosimilar) (N=350) | Lucentis (Ranibizumab) (N=354)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 3 (4) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 2 (3) | 1 (1)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 1 (1) | 1 (1)
Retinal pigment epithelial tear (Eye disorders) | 1 (1) | 0 (0)
Subretinal fluid (Eye disorders) | 1 (1) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vitritis (Eye disorders) | 1 (1) | 0 (0)
Cataract subcapsular (Eye disorders) | 0 (0) | 1 (1)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 2 (2)
Retinal artery occlusion (Eye disorders) | 0 (0) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bacterial colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral circulatory failure (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB11 (Proposed Ranibizumab Biosimilar) (N=350) | Lucentis (Ranibizumab) (N=354)
Neovascular age-related macular degeneration (Eye disorders) | 26 (26) | 24 (24)
Visual acuity reduced (Eye disorders) | 21 (27) | 23 (31)
Conjunctival haemorrhage (Eye disorders) | 19 (23) | 19 (21)
Nasopharyngitis (Infections and infestations) | 39 (44) | 36 (41)
Intraocular pressure increased (Investigations) | 24 (47) | 29 (77)
Hypertension (Vascular disorders) | 17 (18) | 28 (39)

LIMITATIONS AND CAVEATS:
Investigator agree to submit any proposed publication/presentation to Sponsor for review at least sixty days prior to submitting any such proposed publication to a publisher or proceeding with such proposed presentation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT03150589/Prot_SAP_000.pdf